CLINICAL TRIAL: NCT06318494
Title: Analysis of Jumping in Patients With Ankle Instability (Ankle-optogait)
Acronym: Ankle-optoga
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Ankle-optogait
Record Dates: First submitted 2024-03-04; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Ankle Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients suffering from ankle instability (Experimental)
  Interventions: Other: jumping performance
- Healthy volunteer subjects not affected by ankle pathology (Active Comparator)
  Interventions: Other: jumping performance

INTERVENTIONS:
Other: jumping performance — Patients suffering from chronic ankle instability symptomatic of recurrent subjective and objective instability will be considered. Patients will be compared to a control group of healthy volunteer subjects.
  T0 Explanation of the study and written informed consent.
  * Verification of inclusion/exclusion criteria and verification of previous or ongoing treatments.
  * AOFAS Rating Scales,
  * Tegner activity level
  * Vertical Jump Test (CMJ) by foot pedal

SUMMARY:
The study is, in accordance with current legislation, definable as a single-center interventional study with evaluations carried out at a single timeframe.

The objective of the study is to compare jumping performance between subjects with ankle instability and healthy volunteer subjects.

In particular, the primary objective is to verify the difference in the monopodalic CMJ value of the diseased limb of subjects with ankle instability compared to the control group at time 0.

The population is made up of patients suffering from ankle instability and a control group of healthy volunteers, divided as follows:

25 subjects GROUP A: Study group: patients suffering from ankle instability

25 subjects GROUP B: control group: healthy voluntary subjects not affected by ankle pathology

DETAILED DESCRIPTION:
Ankle sprains are one of the most common injuries during sports activity which often results in chronic instability of the ankle, characterized by a feeling of sagging more or less associated with pain with impairment of sports activity.

Numerous authors have suggested that there is altered peripheral neuromuscular control in patients with ankle instability with limitations related to proprioception, neuromuscular control, or strength, leading to deficits not only of the ankle joint but of the entire inferior kinetic chain Jumping is a simple gesture, present in almost every sporting activity, and its evaluation has proven to be a reliable parameter in terms of partisan capacity.

Patients suffering from chronic ankle instability symptomatic of recurrent subjective and objective instability will be considered. Patients will be compared to a control group of healthy volunteer subjects.

T0

* Explanation of the study and written informed consent.
* Verification of inclusion/exclusion criteria and verification of previous or ongoing treatments.
* AOFAS Rating Scales,
* Tegner activity level
* Vertical Jump Test (CMJ) using OptoGait platform using a battery of monopodalic jumps.
* Drop jump using an OptoGait platform using a battery of monopodalic jumps
* Side hop test using an OptoGait platform using a battery of monopod jumps

ELIGIBILITY:
Inclusion Criteria:

* Athletes of legal age (aged between 18 and 45 years inclusive) suffering from chronic ankle instability symptomatic of recurrent subjective and objective instability (study group).
* Athletes of legal age (aged between 18 and 45 years) who are not symptomatic for ankle diseases (control group)
* Signing of the Informed Consent and consent to collaborate in all study procedures.

Exclusion Criteria:

* Minors
* Pregnant women (self-declaration)
* patients with BMI ≥ 30
* patients with orthopaedic, muscular and neuromuscular problems at the time of performing the jump
* Non-acceptance of informed consent
* Patients with previous unilateral or contralateral ankle reconstructive surgery

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
verify the difference in the monopodalic CMJ (countermovement jump test) of the diseased limb of subjects with ankle instability compared to the control group | Day 0
  verify the difference in the monopodalic CMJ (countermovement jump test) value of the diseased limb of subjects with ankle instability compared to the control group at time 0

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico San Siro, Milan, Italy

IPD SHARING:
Plan to Share IPD: No